CLINICAL TRIAL: NCT03193606
Title: Radiographic Assessment of Glass Ionomer Restorations With and Without Prior Application of Nano Silver Fluoride in Occlusal Carious Molars Treated With Partial Caries Removal Technique (Randomized Clinical Trial)
Brief Title: Radiographic Assessment of Glass Ionomer Restorations With and Without Prior Application of Nano Silver Fluoride in Occlusal Carious Molars Treated With Partial Caries Removal Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rahma Ahmed Ibrahem Hafiz, teaching assisstant, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-06-15
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Partial Dentin Caries Removal

STUDY DESIGN:
Intervention Model Description: split mouth randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nano silver fluoride solution (Experimental): carious dentin to be treated with partial caries excavation with application of nano silver fluoride solution prior to glass ionomer restoration.
  Interventions: Other: nano silver fluoride solution
- no nano silver fluoride (No Intervention): carious dentin to be treated with partial caries excavation without application of nano silver fluoride solution restored directly with glass ionomer.

INTERVENTIONS:
Other: nano silver fluoride solution — prepared Nano-silver fluoride could have the capability to arrest caries. As its Nano silver particles have an antimicrobial activity against Mutans Streptococci and Lactobacilli; the main pathogens involved in the development of carious lesions. In addition, its fluoride component is well known to enhance remineralization and inhibit bacterial activity. So, Nano silver fluoride could be a promising solution to combat residual bacteria in tooth cavity with effective remineralization potential on remaining carious dentin
  Arms: nano silver fluoride solution

SUMMARY:
eligible teeth will be randomly divided into two groups to be treated with incomplete caries excavation (A), where (A1) represents teeth to be treated with application of Nano silver fluoride solution on remaining carious dentin prior to final permanent glass ionomer restoration application, (A2) represents comparator group to be restored without Nano silver fluoride application prior to restoration. Every participant will receive both the intervention and control treatment. Image of radiographic density of remaining carious dentin will be evaluated using PSP plate at baseline immediately after restoration and after 6 months after restorative procedures.

The null hypothesis tested is that application of Nano silver fluoride solution prior to glass ionomer restoration will not increase radiopacity of the underlying dentin treated by incomplete carious removal technique compared to that of direct glass ionomer restoration without prior application of Nano silver fluoride.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with at least 2 teeth with active carious lesions limited to the occlusal surface of molars at risk of pulp exposure during direct complete excavation (primary caries lesion involving more than half of the entire dentin thickness determined radiographically).
* Signs and symptoms indicative of pulp vitality, i.e. a positive response to thermal stimulation during a cold test
* Absence of apical pathosis, clinical diagnosis of pulp exposure, fistula, swelling of periodontal tissues.

Exclusion Criteria:

* Teeth with spontaneous pain or sensitivity to percussion.
* Teeth with periodontal lesions, internal or external root resorption, mobility of tooth, sinus opening, or abscessed tooth.
* Radiographic examination revealed, interrupted or broken lamina dura, widened periodontal ligament space, periapical radiolucency.
* patients with systemic medical conditions
* pregnant females

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Caries remineralization. (Mineral density) | six months
  using Density measurement tool in the Digora software

SECONDARY OUTCOMES:
dentin bridge formation. | six months
  Linear measurement tool in the Digora software in Mm

CONTACTS AND LOCATIONS:
Overall Officials: Heba Ah El deeb, Study Director — Associate professor, Conservative dentistry department Cairo University
Locations (1):
- Rahma Ahmed, Giza, Egypt

REFERENCES:
- [Background] Santos VE Jr, Vasconcelos Filho A, Targino AG, Flores MA, Galembeck A, Caldas AF Jr, Rosenblatt A. A new "silver-bullet" to treat caries in children--nano silver fluoride: a randomised clinical trial. J Dent. 2014 Aug;42(8):945-51. doi: 10.1016/j.jdent.2014.05.017. Epub 2014 Jun 12. PMID 24930870